CLINICAL TRIAL: NCT05144178
Title: Insight Into the UAE Experience With Monoclonal Antibodies (Sotrovimab ) as Part of Emirats Health Service (EHS)Fighting Strategy Against COVID-19.
Brief Title: Insight Into the UAE Experience With Monoclonal Antibodies (Sotrovimab )
Acronym: EHS-Strategy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emirates Health Services (EHS) (Other Government)
Responsible Party: Principal Investigator, Dr. Sumaya Abdalateef, Clinical Director, Emirates Health Services (EHS)
Other Study IDs: No.108/ 2021.EHS
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Respiratory Infection
Keywords: Sotrovimab; UAE experience; Emirates health service EHS strategy; Out patient treatment for COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild and moderated COVID -19 patient treated out side the hospital sitting: Reviewing files of such group that had been received Sotrovimab

SUMMARY:
Sotrovimab is a newly developed monoclonal antibody for the treatment of mild and moderate COVID-19 patient, who are at high risk for progression to severe COVID-19, including hospitalization or death. This includes, for example, individuals who are 65 years of age and older or individuals who have certain medical conditions.

The safety and effectiveness of this investigational therapy continues to be evaluated for treatment of COVID-19. Sotrovimab is not authorized for patients who are hospitalized due to COVID-19 or require oxygen therapy due to COVID-19.

As the clinical trial results are too preliminary for the drug to enter routine use in UAE the drug approved only for emergency use, until further evidence shows Sotrovimab is effective, so we thought about this study as a tool to assess the success of Emirats Health service (EHS) strategy for fighting against COVID-19 outside the hospital setting.

DETAILED DESCRIPTION:
May 26, 2021, the U.S. Food and Drug Administration issued an emergency use authorization (EUA) for the treatment of mild-to-moderate coronavirus disease 2019 (COVID-19), as described in the Scope of Authorization (Section II) of this letter, pursuant to Section 564 of the Federal Food, Drug, and Cosmetic Act (the Act) (21 U.S.C. §360bbb-3).

May 28,2021 the UAE Ministry of Health and Prevention approved the investigational drug for emergency use, and Emirats health service considered strategy for fighting against COVID-19 outside the hospital setting, based on this strategy ,special protocol was finalized and approved including initiation of infusion units for the drug in EHS hospital and primary health care centers, all Infection Prevention and Control Precautions were taken inconsideration .

The overall aim of this study is to determine the effectiveness of Sotrovimab infusion in cohort of ambulatory patients with early symptomatic COVID-19 at high risk for hospitalization, in UAE. We expect to assess the Proportion of patients who have progression of COVID-19 through 28 days as defined by visit to a hospital emergency room for management or illness, or hospitalization more than 24 h for acute management of illness or death. files of patients treated from June 2021 till October 2021 will be reviewed and data will be collected based on the protocol approved from MOHAP ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* All cases received Sotrovimab according the EUA protocol.
* All patient aged 13 and above

Exclusion Criteria:

* Sever form of the COVID-19 disease
* Hospitalized patient
* Age less than 13 years old
* BMI less than 25 and no risk factors

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The source population will consist of individuals residing in UAE ,infected with SARS-CoV-2 and developed mild or moderate symptoms and are high risk .
  High risk patients are defined as meeting at least 1 of the following criteria:
  1. BMI ≥ 25
  2. Chronic kidney disease
  3. Diabetes
  4. Immunosuppressive disease
  5. Receiving immunosuppressive treatment
  6. Age ≥ 65 years
  7. Age ≥ 55 years and have cardiovascular disease, hypertension, or COPD/chronic respiratory disease.
  8. pregnancy
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2021-11-14 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-09 (Estimated)

PRIMARY OUTCOMES:
percent of hospital admission from total number of reviewed patient | 10 days
  Admission to hospital with progressive COVID -19 more than 24h
percent of Death among total number of reviewed patient | 28 days
  mortality post treatment

CONTACTS AND LOCATIONS:
Overall Officials: sumaya abdalateef, Principal Investigator — Emirats Health Service (EHS)
Locations (1):
- Emirats Health Service, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided